CLINICAL TRIAL: NCT00101803
Title: Efficacy and Safety of Vildagliptin in Combination With Pioglitazone in Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2355
Record Dates: First submitted 2005-01-13; First posted 2005-01-14 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
Many people with type 2 diabetes cannot maintain target blood glucose levels when taking a single oral drug. The purpose of this study is to assess the safety and effectiveness of the combination of vildagliptin, an unapproved drug, and pioglitazone in lowering overall blood glucose levels in people with type 2 diabetes who have not previously been treated with drug therapy to lower their blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Not previously treated with oral antidiabetic agents as defined by the protocol
* Blood glucose criteria must be met
* Body mass index (BMI) in the range 22-45

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes
* Evidence of serious diabetic complications
* Evidence of serious cardiovascular complications
* Laboratory value abnormalities as defined by the protocol
* Known sensitivity to pioglitazone
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2005-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose at 24 weeks
Adverse event profile after 24 weeks of treatment
Patients with endpoint HbA1c <7% after 24 weeks
Patients with endpoint HbA1C <6.5% after 24 weeks
Patients with reduction in HbA1c >/= to 0.7% after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Pratley RE, Schweizer A, Rosenstock J, Foley JE, Banerji MA, Pi-Sunyer FX, Mills D, Dejager S. Robust improvements in fasting and prandial measures of beta-cell function with vildagliptin in drug-naive patients: analysis of pooled vildagliptin monotherapy database. Diabetes Obes Metab. 2008 Sep;10(10):931-8. doi: 10.1111/j.1463-1326.2007.00835.x. Epub 2007 Dec 17. PMID 18093207
- [Derived] Pratley RE, Rosenstock J, Pi-Sunyer FX, Banerji MA, Schweizer A, Couturier A, Dejager S. Management of type 2 diabetes in treatment-naive elderly patients: benefits and risks of vildagliptin monotherapy. Diabetes Care. 2007 Dec;30(12):3017-22. doi: 10.2337/dc07-1188. Epub 2007 Sep 18. PMID 17878242
- [Derived] Rosenstock J, Kim SW, Baron MA, Camisasca RP, Cressier F, Couturier A, Dejager S. Efficacy and tolerability of initial combination therapy with vildagliptin and pioglitazone compared with component monotherapy in patients with type 2 diabetes. Diabetes Obes Metab. 2007 Mar;9(2):175-85. doi: 10.1111/j.1463-1326.2006.00698.x. PMID 17300593